CLINICAL TRIAL: NCT04383431
Title: Standard Cross-linking Versus Accelerated Photoactivated Chromophore Cross-linking (PACK-CXL) for Treatment of Infectious Keratitis: A Comparative Study
Brief Title: Cross-linking as Treatment in Infectious Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Assistant Professor of Ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-9/12/2018
Record Dates: First submitted 2020-04-27; First posted 2020-05-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Infectious Keratitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard CXL (Experimental): Standard epithelium-off CXL, 30 minutes soaking time with riboflavin, 30 minutes UVA corneal irradiation continuous mode.
  Interventions: Procedure: PACK-CXL
- Accelerated CXL (Experimental): Accelerated epithelium-off CXL, 12 minutes soaking time with riboflavin, 8 minutes UVA corneal irradiation continuous mode.
  Interventions: Procedure: PACK-CXL

INTERVENTIONS:
Procedure: PACK-CXL — Standard epithelium-off CXL, 12 minutes soaking time with riboflavin, 8 minutes UVA corneal irradiation pulsed mode.

SUMMARY:
To compare between SCXL and ACXL for treatment of infectious keratitis

DETAILED DESCRIPTION:
Standard epithelium-off CXL, 30 minutes soaking time with riboflavin, 30 minutes UVA corneal irradiation continuous mode (Group A). Accelerated CXL 11 minutes soaking time with riboflavin, 8 minutes UVA corneal irradiation pulsed mode (Group B).

ELIGIBILITY:
Inclusion Criteria:

* Fungal infectious keratitis
* bacterial infectious keratitis
* Must be not responding to medication

Exclusion Criteria:

* Viral keratitis
* Pregnancy and lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Corneal healing | 3 months
  Reepithelization of corneal ulcer which is measured in mm by slitlamp examination
Corneal edema | 3 months
  measurement of corneal edema by measurement of the corneal thickness in um by Optical Coherent Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal, MD. PhP, Principal Investigator — 00201068559840
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be allowed for sharing
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months after end of study
Access Criteria: Ophthalmologists are allowed for access of data. they should email the principal investigator via dr_m_iqbal@yahoo.com to get the permission after reviewing the qualifications and quality of request